## UNIVERSITI MALAYA MEDICAL CENTRE

CONSENT BY PATIENT FOR CLINICAL RESEARCH

Version Date: 22<sup>nd</sup> March 2023

| I, | ) |
|---|---|
| of | |
| (Address) hereby agree to take part in the clinical research (clinical study) specified below: | |
| <u>Title of Study:</u> Efficacy and Health Economics of Antimicrobial-impregnated Central Venous Catheters (CVCs) compared to Non-impregnated CVCs in Central Line-associated Bloodstream Infection (CLABSI) Prevention in a Malaysia University Hospital Adult Intensive Care Unit (ICU) | |
| the nature and purpose of which has been explained to me by | |
| Dr | (Name & Designation of Interpreter) |
| to the best of his/her ability in language/dia | lect. |
| I have been told about the nature of the clinical research in terms of methodology, possible adverse effects and complications (as per patient information sheet). After knowing and understanding all the possible advantages and disadvantages of this clinical research, I voluntarily consent of my own free will to participate in the clinical research specified above. | |
| I understand that I can withdraw from this clinical research at any time without assigning any reason whatsoever and in such a situation shall not be denied the benefits of usual treatment by the attending doctors. | |
| Date: Signature or Thumbprint (Patient) IN THE PRESENCE OF | |
| Name | Signature (Witness for Signature of Patient) ove-mentioned clinical research. |
| Date Signature | (Attending Doctor) |

R.N. **CONSENT BY PATIENT** Name **FOR** Sex **CLINICAL RESEARCH** Age

Unit

## UNIVERSITI MALAYA MEDICAL CENTRE

Version No.: 1

**Version Date: 22<sup>nd</sup> March 2023** 

## CONSENT BY RESPONSIBLE RELATIVE FOR CLINICAL RESEARCH

| I. | Identity Card No |
|---|---|
| (Name) | |
| (Address) | |
| | Identity Card No |
| (Name) participate in the clinical research (clinical study) specified by | below:- |
| | microbial-impregnated Central Venous Catheters (CVCs) sociated Bloodstream Infection (CLABSI) Prevention in a (ICU) |
| the nature and purpose of which has been explained to me by | у |
| Dr and inte | rpreted by(Name & Designation of Interpreter) |
| to the best of his/her ability in | language/dialect. |
| | terms of procedure, possible adverse effects and complications advantages and disadvantages of participating in this research. n this research specified above. |
| I understand that I can withdraw my relative from this clinical research at any time without assigning any reason whatsoever and in such situation, my relative shall not be denied the benefits of usual treatment by the attending doctors. Should my relative regains his/her ability to consent, he/she will have the right to remain in this research or may choose to withdraw. | |
| Relationship | Signature or |
| Date: to Patient | Thumbprint |
| IN THE PR | RESENCE OF |
| Name | Signature<br>(Witness) |
| I confirm that I have explained to the patient's relative the nature and purpose of the above-mentioned clinical research. | |
| Date | Signature(Attending Doctor) |

CONSENT BY
RESPONSIBLE RELATIVE FOR
CLINICAL RESEARCH

R.N. Name Sex Age Unit